CLINICAL TRIAL: NCT05122988
Title: Facing Adverse Childhood Experiences Using New Technologies
Brief Title: Facing Adverse Childhood Experiences
Acronym: FACE
Status: Completed | Type: Observational
Sponsor: University of Applied Sciences and Arts Northwestern Switzerland (Other)
Responsible Party: Principal Investigator, Jeannette Brodbeck, Prof. Dr., University of Applied Sciences and Arts Northwestern Switzerland
Other Study IDs: SNF Nr. 100019_197731
Record Dates: First submitted 2021-09-27; First posted 2021-11-17 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Adverse Childhood Experiences
Keywords: Adverse childhood experiences; psychosocial functioning; emotion regulation; social information processing; social support
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- age 18: n=1017
- age 19: n=676
- age 20: n=337
- age 21: n=500

SUMMARY:
Childhood experiences affect psychosocial well-being and mental health across the life course for better or worse. The aim of the present study is to investigate how adverse childhood experiences before the age of 18 impact psychological functioning in young adulthood, and whether social information processing and emotion regulation may mediate these associations.

DETAILED DESCRIPTION:
The study plans to recruit 5000 young adults aged 18 to 21 representative of the German speaking Swiss population. Participant will be invited to the study by mail. Addresses stem from a Swiss sampling registry ("Stichprobenregister SRPH") and are provided by the Swiss Statistical Office. Access to this address lists is reserved to studies of national interest that are funded by the Swiss National Science foundation. Data collection will be conducted online with a REDCap survey following an accelerated cohort design. After the baseline measurement (w1), three follow ups are planned after 1 year (w2), 2 years (w3) and 3 years (w4), resulting in ages 18 to 24 being covered. The primary outcome will be psychosocial functioning across the study period.

1. Primary objective:

   The primary objective of the study is to analyse the longitudinal associations between childhood experiences, emotion regulation, social information processing, social support and psychosocial functioning in young adults.
   * Hypothese 1 is that adverse childhood experiences (ACE) are associated with a higher risk for lower psychosocial functioning in young adulthood and 2) that this association is mediated by deficits in emotion regulation, social information processing and lower social support.
   * Hypothese 2 is that positive childhood experiences are associated with higher social support, adaptive emotion regulation and high well-being in young adulthood and that good relationships with parents and high social support are a protective factor in the presence of adversities.
   * Hypothese 3 is that among young adults with ACE, higher social support, seeking professional help and more adaptive coping strategies are associated with a more adaptive psychosocial functioning.

   Secondary objectives are
2. to examine the effect of childhood experiences on emotion regulation and social information processing.
3. to investigate the effects of emotion regulation and social information processing on the quality of friendships and social support.
4. to analyse the longitudinal associations of childhood experiences, emotion regulation, social information processing, social support and the single variables that constitute the composite score of psychosocial functioning, e.g. well-being, psychosocial distress, risk behaviours.
5. to investigate the associations between ACE, emotion regulation and social information processing and seeking professional support.
6. Further exploratory hypotheses investigate whether there are patterns of ACE which show differential associations with emotion regulation, social information processing, support and psychosocial functioning or single variables of psychosocial functioning.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 21, Living in German-speaking Switzerland, Internet Access

Exclusion Criteria:

* Insufficient mastery of German

Ages: 18 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: General population of 18 to 21 years old from the German speaking region of Switzerland. Adresses stem from the Swiss household survey and are provided by the Federal Statistical Office.
Sampling Method: Probability Sample
Enrollment: 2606 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Latent composite score for psychosocial functioning | a baseline measurement (w1)
  A single latent score for overall psychosocial functioning will be created out of the following individual variables using the MPlus software: Well-being (Ryff & Keyes 1995), Internalizing (Spitzer et al., 2011) and externalizing (Renshaw & Cook 2019) psychopathological symptoms, psychosocial burden (Brodbeck et al., 2007) and functioning in social und and work situations (Mundt et al., 2002). A higher score indicates better overall psychological functioning.
Latent composite score for psychosocial functioning | change over 3 years (from w1 to w4)
  A single latent score for overall psychosocial functioning will be created out of the following individual variables using the MPlus software: Well-being (Ryff & Keyes 1995), Internalizing (Spitzer et al., 2011) and externalizing (Renshaw & Cook 2019) psychopathological symptoms, psychosocial burden (Brodbeck et al., 2007) and functioning in social und and work situations (Mundt et al., 2002). A higher score indicates better overall psychological functioning.
Psychological Well-being | a baseline measurement (w1)
  Six dimensions (autonomy, environmental mastery, personal growth, positive relations with others, purpose in life, and self-acceptance) measured with Ryffs Well-being scale (Ryff & Keyes 1995), 42 item Version (Abbott et al., 2010). Scores for the subscales range from 7 to 42, and scores for the total scale from 42 to 294. A higher score indicates better well-being.
Psychological Well-being | change over 3 years (from w1 to w4)
  Six dimensions (autonomy, environmental mastery, personal growth, positive relations with others, purpose in life, and self-acceptance) measured with Ryffs Well-being scale (Ryff & Keyes 1995), 42 item Version (Abbott et al., 2010). Scores for the subscales range from 7 to 42, and scores for the total scale from 42 to 294. A higher score indicates better well-being.
Internalizing symptoms | a baseline measurement (w1)
  Measured with the 18-item Brief Symptom Inventory (BSI-18) (Spitzer et al., 2011), containing questions about depressivity, anxiety and somatic symptoms. The total score ranges from 18 to 90, and a higher score indicates more internalizing symptoms.
Internalizing symptoms | change over 3 years (from w1 to w4)
  Measured with the 18-item Brief Symptom Inventory (BSI-18) (Spitzer et al., 2011), containing questions about depressivity, anxiety and somatic symptoms. The total score ranges from 18 to 90, and a higher score indicates more internalizing symptoms.
Externalizing symptoms | a baseline measurement (w1)
  Measured with the 10-item Externalizing Problems Screener (Renshaw & Cook 2019). Total score ranges from 0 to 40, with a higher score indicating more externalizing symptoms.
Externalizing symptoms | change over 3 years (from w1 to w4)
  Measured with the 10-item Externalizing Problems Screener (Renshaw & Cook 2019). Total score ranges from 0 to 40, with a higher score indicating more externalizing symptoms.
Functioning in social und and work situations | a baseline measurement (w1)
  Measured with the 5-item Work and Social Adjustment Scale (Mundt et al., 2002), measuring impairment in different social and work situations. The total score ranges from 0 to 40, with a higher score indicating worse functioning in social and work situations.
Functioning in social und and work situations | change over 3 years (from w1 to w4)
  Measured with the 5-item Work and Social Adjustment Scale (Mundt et al., 2002), measuring impairment in different social and work situations. The total score ranges from 0 to 40, with a higher score indicating worse functioning in social and work situations.

SECONDARY OUTCOMES:
Help seeking behaviour | a baseline measurement (w1)
  We asked whether participants ever sought professional help due to psychological and social problems. If yes, we asked about whether they sought help in eight different types of support setting (e.g. psychotherapy, general practitioner, psychological service at school).
Help seeking behaviour | change over 3 years (from w1 to w4)
  We asked whether participants ever sought professional help due to psychological and social problems. If yes, we asked about whether they sought help in eight different types of support setting (e.g. psychotherapy, general practitioner, psychological service at school).
Social Support | a baseline measurement (w1)
  Measured with the 14-Item social support scale (Fydrich et al., 2009). The total score ranges from 14 to 70, with a higher score indicating better social support.
Social Support | change over 3 years (from w1 to w4)
  Measured with the 14-Item social support scale (Fydrich et al., 2009). The total score ranges from 14 to 70, with a higher score indicating better social support.
Substance use | a baseline measurement (w1)
  Participants were asked how frequently they used tobacco, alcohol, cannabis, party drugs, cocaine/heroin, other drugs and pharmaceutical drugs for non-medical use. For substances they used, they were additionally asked the age of first use and the 4-item Addiction Screener (Schluter et al., 2018). The total score for the addiction screener ranges from 0 to 16, with a higher score indicating worse outcomes.
Substance use | change over 3 years (from w1 to w4)
  Participants were asked how frequently they used tobacco, alcohol, cannabis, party drugs, cocaine/heroin, other drugs and pharmaceutical drugs for non-medical use. For substances they used, they were additionally asked the age of first use and the 4-item Addiction Screener (Schluter et al., 2018). The total score for the addiction screener ranges from 0 to 16, with a higher score indicating worse outcomes.
Psychosocial Burden | a baseline measurement (w1)
  Participants were asked to which degree they felt burdened in 13 different areas of life, for example school/work, sleep, romantic relationship, physical health, financial situation (Brodbeck et al., 2007). The total score ranges from 0 to 130, with a higher score indicating more burden.
Psychosocial Burden | change over 3 years (from w1 to w4)
  Participants were asked to which degree they felt burdened in 13 different areas of life, for example school/work, sleep, romantic relationship, physical health, financial situation (Brodbeck et al., 2007). The total score ranges from 0 to 130, with a higher score indicating more burden.

OTHER OUTCOMES:
Social information processing: Social Intelligence | a baseline measurement (w1)
  Measured with the 14-item Tromsø Social Intelligence Scale (Silvera et al., 2001). The total score ranges from 14 to 98, with a higher score indicating a higher social intelligence.
Social information processing: Social Intelligence | change over 3 years (from w1 to w4)
  Measured with the 14-item Tromsø Social Intelligence Scale (Silvera et al., 2001). The total score ranges from 14 to 98, with a higher score indicating a higher social intelligence.
Social information processing: Hostile interpretation bias | a baseline measurement (w1)
  Measured with the 32-item Hostile interpretation bias scale (Dillon et al., 2016). The total score for the hostile scale (16 items) ranges from 0 to 96, with a higher score indicating a more hostile interpretation.
Social information processing: Hostile interpretation bias | change over 3 years (from w1 to w4)
  Measured with the 32-item Hostile interpretation bias scale (Dillon et al., 2016). The total score for the hostile scale (16 items) ranges from 0 to 96, with a higher score indicating a more hostile interpretation.
Social information processing: Rejection sensitivity | a baseline measurement (w1)
  Measured with the 18-item Rejection sensitivity questionnaire (Berenson et al., 2009). The total score ranges from 9 to 54, with a higher score indicating a higher rejection sensitivity.
Social information processing: Rejection sensitivity | change over 3 years (from w1 to w4)
  Measured with the 18-item Rejection sensitivity questionnaire (Berenson et al., 2009). The total score ranges from 9 to 54, with a higher score indicating a higher rejection sensitivity.
Emotion regulation: Perseverative Thinking | a baseline measurement (w1)
  Measured with the 15-item Perseverative Thinking Questionnaire (Ehring et al., 2011).The total score ranges from 0 to 60, with a higher score indicating more preservative thinking.
Emotion regulation: Perseverative Thinking | change over 3 years (from w1 to w4)
  Measured with the 15-item Perseverative Thinking Questionnaire (Ehring et al., 2011).The total score ranges from 0 to 60, with a higher score indicating more preservative thinking.
Emotion regulation: Emotion Reactivity | a baseline measurement (w1)
  Measured with the 21-item Emotion Reactivity Scale (Nock et al., 2008). The total score ranges from 0 to 84, with a higher score indicating a higher emotional reactivity.
Emotion regulation: Emotion Reactivity | change over 3 years (from w1 to w4)
  Measured with the 21-item Emotion Reactivity Scale (Nock et al., 2008). The total score ranges from 0 to 84, with a higher score indicating a higher emotional reactivity.
Emotion regulation: Self-Efficacy for Managing Emotions | a baseline measurement (w1)
  Measured with the 7-item Self-Efficacy for Managing Emotions scale (PROMIS; https://www.healthmeasures.net/explore-measurement-systems/promis). The total score ranges from 7 to 49, with a higher score indicating a better self-efficacy for managing emotions.
Emotion regulation: Self-Efficacy for Managing Emotions | change over 3 years (from w1 to w4)
  Measured with the 7-item Self-Efficacy for Managing Emotions scale (PROMIS; https://www.healthmeasures.net/explore-measurement-systems/promis). The total score ranges from 7 to 49, with a higher score indicating a better self-efficacy for managing emotions.

CONTACTS AND LOCATIONS:
Overall Officials: Jeannette Brodbeck, PHD, Principal Investigator — University of Applied Sciences Northwestern Switzerland
Locations (1):
- University of Applied Science Northwestern Switzerland, Olten, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be available on request to interested researchers
Supporting Information: Study Protocol
Time Frame: After the end of data collection (2025)
Access Criteria: Access to these data is permitted for scientific purposes on request. A data access agreement will be signed and the source of the data (including the funding agency) needs to be acknowledged.

REFERENCES:
- [Background] Bernstein DP, Stein JA, Newcomb MD, Walker E, Pogge D, Ahluvalia T, Stokes J, Handelsman L, Medrano M, Desmond D, Zule W. Development and validation of a brief screening version of the Childhood Trauma Questionnaire. Child Abuse Negl. 2003 Feb;27(2):169-90. doi: 10.1016/s0145-2134(02)00541-0. PMID 12615092
- [Background] Norman RE, Byambaa M, De R, Butchart A, Scott J, Vos T. The long-term health consequences of child physical abuse, emotional abuse, and neglect: a systematic review and meta-analysis. PLoS Med. 2012;9(11):e1001349. doi: 10.1371/journal.pmed.1001349. Epub 2012 Nov 27. PMID 23209385
- [Background] Weissman DG, Bitran D, Miller AB, Schaefer JD, Sheridan MA, McLaughlin KA. Difficulties with emotion regulation as a transdiagnostic mechanism linking child maltreatment with the emergence of psychopathology. Dev Psychopathol. 2019 Aug;31(3):899-915. doi: 10.1017/S0954579419000348. Epub 2019 Apr 8. PMID 30957738
- [Background] Pollak SD. Multilevel developmental approaches to understanding the effects of child maltreatment: Recent advances and future challenges. Dev Psychopathol. 2015 Nov;27(4 Pt 2):1387-97. doi: 10.1017/S0954579415000826. PMID 26535932
- [Background] Abbott RA, Ploubidis GB, Huppert FA, Kuh D, Croudace TJ. An Evaluation of the Precision of Measurement of Ryff's Psychological Well-Being Scales in a Population Sample. Soc Indic Res. 2010 Jul;97(3):357-373. doi: 10.1007/s11205-009-9506-x. Epub 2009 Sep 1. PMID 20543875
- [Background] Berenson KR, Gyurak A, Ayduk O, Downey G, Garner MJ, Mogg K, Bradley BP, Pine DS. Rejection sensitivity and disruption of attention by social threat cues. J Res Pers. 2009 Dec 1;43(6):1064-1072. doi: 10.1016/j.jrp.2009.07.007. PMID 20160869
- [Background] Brodbeck J, Matter M, Page J, Moggi F. Motives for cannabis use as a moderator variable of distress among young adults. Addict Behav. 2007 Aug;32(8):1537-45. doi: 10.1016/j.addbeh.2006.11.012. Epub 2006 Dec 18. PMID 17178197
- [Background] Dillon KH, Allan NP, Cougle JR, Fincham FD. Measuring Hostile Interpretation Bias: The WSAP-Hostility Scale. Assessment. 2016 Dec;23(6):707-719. doi: 10.1177/1073191115599052. Epub 2015 Aug 6. PMID 26251297
- [Background] Ehring T, Zetsche U, Weidacker K, Wahl K, Schonfeld S, Ehlers A. The Perseverative Thinking Questionnaire (PTQ): validation of a content-independent measure of repetitive negative thinking. J Behav Ther Exp Psychiatry. 2011 Jun;42(2):225-32. doi: 10.1016/j.jbtep.2010.12.003. Epub 2010 Dec 21. PMID 21315886
- [Background] Ryff CD, Keyes CL. The structure of psychological well-being revisited. J Pers Soc Psychol. 1995 Oct;69(4):719-27. doi: 10.1037//0022-3514.69.4.719. PMID 7473027
- [Background] Nock MK, Wedig MM, Holmberg EB, Hooley JM. The emotion reactivity scale: development, evaluation, and relation to self-injurious thoughts and behaviors. Behav Ther. 2008 Jun;39(2):107-16. doi: 10.1016/j.beth.2007.05.005. Epub 2007 Oct 29. PMID 18502244
- [Background] Mundt JC, Marks IM, Shear MK, Greist JH. The Work and Social Adjustment Scale: a simple measure of impairment in functioning. Br J Psychiatry. 2002 May;180:461-4. doi: 10.1192/bjp.180.5.461. PMID 11983645
- [Background] Silvera DH, Martinussen M, Dahl TI. The Tromso Social Intelligence Scale, a self-report measure of social intelligence. Scand J Psychol. 2001 Sep;42(4):313-9. doi: 10.1111/1467-9450.00242. PMID 11547906
- [Background] Schluter MG, Hodgins DC, Wolfe J, Wild TC. Can one simple questionnaire assess substance-related and behavioural addiction problems? Results of a proposed new screener for community epidemiology. Addiction. 2018 Aug;113(8):1528-1537. doi: 10.1111/add.14166. Epub 2018 Feb 26. PMID 29357188
- [Background] Spitzer C, Hammer S, Lowe B, Grabe HJ, Barnow S, Rose M, Wingenfeld K, Freyberger HJ, Franke GH. [The short version of the Brief Symptom Inventory (BSI -18): preliminary psychometric properties of the German translation]. Fortschr Neurol Psychiatr. 2011 Sep;79(9):517-23. doi: 10.1055/s-0031-1281602. Epub 2011 Aug 25. German. PMID 21870312
- [Derived] Brodbeck J, Botschi SIR, Vetsch N, Berger T, Schmidt SJ, Marmet S. Investigating emotion regulation and social information processing as mechanisms linking adverse childhood experiences with psychosocial functioning in young swiss adults: the FACE epidemiological accelerated cohort study. BMC Psychol. 2022 Apr 11;10(1):99. doi: 10.1186/s40359-022-00798-5. PMID 35410310